CLINICAL TRIAL: NCT02893124
Title: The Optimizing Treatment of Peginterferon Alpha in HBeAg-negative Chronic Hepatitis B Virus Patients With Low Level HBsAg
Brief Title: The Optimizing Treatment of Peginterferon (PEG IFN) Alpha in Chronic Hepatitis B Virus Patients With Low Level HBsAg
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Peking University (Other); Huazhong University of Science and Technology (Other); Nanchang University (Other); Huizhou Municipal Central Hospital (Other); First People's Hospital, Shunde China (Other); Shenzhen Third People's Hospital (Other); First People's Hospital of Foshan (Other); Tang-Du Hospital (Other); First Affiliated Hospital of Kunming Medical University (Other); Yuebei People's Hospital (Other)
Responsible Party: Principal Investigator, Zhiliang Gao, Chief director of department of infectious disease, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I-Cure-3
Record Dates: First submitted 2016-08-28; First posted 2016-09-08 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Chronic Hepatitis B
Keywords: chronic hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEG-IFN group (Experimental): HBeAg-negative CHB patients with HBsAg <1000 IU/ mL and HBV DNA<100 IU/mL are to receive peginterferon alfa-2a 180 micrograms/week or peginterferon alfa-2b 80 micrograms/week for at most 96 weeks.
  Interventions: Drug: peginterferon alfa
- NAs group (No Intervention): CHB patients do not need to change their NAs treatment.

INTERVENTIONS:
Drug: peginterferon alfa — peginterferon alfa-2a 180 micrograms/week or peginterferon alfa-2b 80 micrograms/week, for at most 96 weeks.
  Other Names: peginterferon alfa-2a or peginterferon alfa-2b
  Arms: PEG-IFN group

SUMMARY:
HBeAg-negative chronic hepatitis B (CHB) patients with low Level HBsAg and with a history of drug resistance or suboptimal/partial virological response were enrolled. After giving informed consent, patients were treated with nucleoside analog(s) (NAs) once a day and weekly subcutaneous injections of alfa-2a 180 micrograms/week or peginterferon alfa-2b 80 micrograms/week for 12 weeks. 12 weeks later, NAs was stopped, patients were treated with weekly subcutaneous injections of alfa-2a 180 micrograms/week or peginterferon alfa-2b 80 micrograms/week. Treatment endpoint was HBsAg loss(<0.05 IU/mL).

DETAILED DESCRIPTION:
It is estimated that more than 400 million people are infected with hepatitis B virus (HBV) globally. HBeAg-negative CHB patients with low Level HBsAg and with a history of drug resistance or suboptimal/partial virological response were enrolled in the out-patient department of 3rd Affiliated Hospital of Sun Yat-sen University. All of them were HBsAg positive and anti-HBs negative for more than 6 months with HBV DNA<100 IU/mL and HBsAg levels <1000 IU/mL. All patients did not have other liver diseases and contraindications for interferon therapy.

After giving informed consent, patients were treated with NAs once a day and weekly subcutaneous injections of alfa-2a 180 micrograms/week or peginterferon alfa-2b 80 micrograms/week for 12 weeks. 12 weeks later, NAs was stopped, patients were treated with weekly subcutaneous injections of alfa-2a 180 micrograms/week or peginterferon alfa-2b 80 micrograms/week. The use of other immune suppressive or regulatory drugs and other antiviral drugs was prohibited during the course of the study.

In this study, treatment endpoint was HBsAg loss(<0.05 IU/mL).Anti-HBs positive(>10 milli-International unit)(mIU/mL) defined as seroconversion. Depending on the decline of HBsAg level, treatment was either continued for a prolonged period (no more than 96 weeks) until the endpoint was achieved, or terminated in case of nonresponse.

ELIGIBILITY:
Inclusion Criteria:

1. CHB patients who had received single NAs for more than 12 months and had a history of NAs drug resistance or suboptimal/partial virological response.
2. Hepatitis B e antigen (HBeAg)-negative.
3. Hepatitis B surface antigen (HBsAg) positive and <1000 IU/mL.
4. Hepatitis B virus DNA <100 IU/mL.

Exclusion Criteria:

1. Patients with liver cirrhosis, Hepatocellular Carcinoma or alpha feto protein (AFP) >2 upper limit of normal(ULN) or other malignancies.
2. Patients with other factors causing liver diseases.
3. Pregnant and lactating women.
4. Patients with concomitant HIV infection or congenital immune deficiency diseases.
5. Patients with diabetes, autoimmune diseases.
6. Patients with important organ dysfunctions.
7. Patients with serious complications (e.g., infection, hepatic encephalopathy, hepatorenal syndrome, gastrointestinal bleeding.)
8. Patients who receive antineoplastic or immunomodulatory therapy in the past 12 months.
9. Patients with a previous use of IFN anti hepatitis B virus treatment.
10. Patients who can't come back to clinic for follow-up on schedule.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
HBsAg Clearance | 96 weeks
  Percentage of Participants with HBsAg <0.05 IU/mL.

SECONDARY OUTCOMES:
HBsAg Seroconversion | 96 weeks
  Percentage of Participants with HBsAg <0.05 IU/mL and anti-HBsAg positive.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Infectious Diseases, The Third Affliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided